CLINICAL TRIAL: NCT03612895
Title: Proactive Population Health Strategy to Offer Tobacco Dependence Treatment to Smokers in a Primary Care Practice Network
Brief Title: Proactive Population Health Strategy to Offer Tobacco Dependence Treatment to Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Nancy A. Rigotti, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015P0021111
Record Dates: First submitted 2018-07-21; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Smoking, Tobacco
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internal Care Coordination (Experimental): The smoker will be connected to a Tobacco Care Coordinator who is based centrally within the health care system but has ready access via EHR, email, and telephone with staff in each primary care practice.
  Interventions: Behavioral: Internal Care Coordination
- External Community Referral (Experimental): This intervention will connect the smoker directly via "warm transfer" to a the Massachusetts Smokers Helpline operated by National Jewish Health, which will provide its standard services to smokers.
  Interventions: Behavioral: External Community Referral
- Usual Care (Other): Passive referral to quitline and referral to primary care physician.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Internal Care Coordination — This individual will primarily initiate, guide, and optimize adherence to the care that others deliver, rather than providing direct care his or herself. S/he will call the smoker to conduct a brief assessment of tobacco use and readiness to quit, offer brief counseling and motivational intervention, describe the available pharmacologic and behavioral options, help the smoker to choose among them, and link the smoker to chosen resources. The resources offered will include both internal (health care system based) and external (community based) tobacco cessation resources.
  Arms: Internal Care Coordination
Behavioral: External Community Referral — Massachusetts (MA) Helpline services include an assessment of smoking history and readiness to quit, advice to quit, self-help materials and telephone counseling. For smokers who set a quit date in the next 30 days, the Helpline offers up to 5 proactive telephone counseling calls with options for text messaging and web-based resources. It also provides eligible smokers 4 weeks of free nicotine patch or gum mailed to their home.
  Arms: External Community Referral
Behavioral: Usual Care — Participants will be given the number to the MA Smokers Helpline and advised to contact their primary care provider for additional assistance in quitting smoking.
  Arms: Usual Care

SUMMARY:
Health care systems are key channels for delivering tobacco cessation treatment to the smokers in a population. A population-based approach could complement office-based care and offload busy clinicians. The project will conduct population-based proactive outreach to current smokers in a health care system's primary care practices and randomize smokers who respond to the outreach to 3 groups: 2 alternative evidence-based cessation resources or to usual care.

Specific Aims:

Aim 1: To determine the feasibility and reach of the program

Aim 2a: To determine whether the 2 intervention arms combined increase the proportion of smokers who use tobacco cessation treatment over a 6-month follow-up compared to those randomized to usual clinical care.

Aim 2b: To determine whether each of the two intervention arms increases the proportion of smokers who use tobacco cessation treatment over a 6-month follow-up, compared to those receiving usual clinical care.

DETAILED DESCRIPTION:
Health care systems are key channels for delivering tobacco cessation treatment to the smokers in a population. Current health care system approaches require busy clinicians with many competing demands on their time to initiate treatment in the course of clinical encounter. A population-based approach is an alternative that could complement office-based care and offload busy clinicians. The ongoing evolution of the health care system is making this more feasible with adoption of electronic health records (EHR) that document patients' smoking status in a coded field. This facilitates the creation of a registry of smokers who can be offered tobacco treatment proactively. However, the optimal way to implement a proactive population health strategy for tobacco users is unclear.

The goal of the project is to implement a population-based proactive outreach program to current smokers in a health care system's primary care practices. The program will

1. Proactively contact smokers independent of their health care visits and
2. Connect smokers who respond to evidence-based tobacco cessation resources available in the health care system and/or community.

The study aims of the study are to:

Aim 1: To determine the feasibility and reach of the program.

Aim 2a: To determine whether the two intervention arms combined increase the proportion of smokers who use tobacco cessation treatment over a 6-month follow-up, compared to those receiving usual clinical care.

Aim 2b: To determine whether each of the two interventions increases the proportion of smokers who use tobacco cessation treatment over a 6-month follow-up, compared to those receiving usual clinical care.

Exploratory aim: To compare the 7-day point prevalence smoking cessation rate in each intervention arm to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Seen at a participating Massachusetts General Hospital (MGH) Primary Care practice within the linkage cohort time period
* "Current Smoker" as reported within the year based upon structured field in the health monitoring section of the electronic health record, or problem list term
* Listed telephone number

Exclusion Criteria:

* Excluded by primary care provider
* No telephone in electronic health record or at primary care provider's office
* Non-English speaking
* Problem list has a diagnosis of dementia, psychosis, schizophrenia, Alzheimer's disease, delirium, schizoaffective disorder, or suicidal tendencies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are provided any evidence-based tobacco cessation treatment (as defined below), comparing pooled intervention groups (Internal Care Coordination + External Community Referral) vs Usual Care | 6 months
  Any tobacco cessation treatment was defined as any of the following: (1) in-person visit with the practice-based tobacco counselor; (2) completion of >1 Quitline counseling call (excluding the initial registration call in which the participant was transferred from the interactive voice response [IVR] system); (3) telephone contact with the study's Tobacco Coach (excluding the initial call after enrollment); (4) outpatient prescription for nicotine replacement, bupropion, or varenicline in the EHR; or (5) provision of nicotine replacement by the Quitline. Information was obtained from the EHR, research program records, practice-based tobacco counselor records, and the Quitline provider, National Jewish Health

SECONDARY OUTCOMES:
Proportion of patients who are provided any evidence-based tobacco cessation treatment (defined below), comparing Internal Care Coordination vs. Usual Care | 6 months
  Any tobacco cessation treatment was defined as any of the following: (1) in-person visit with the practice-based tobacco counselor; (2) completion of >1 Quitline counseling call (excluding the initial registration call in which the participant was transferred from the IVR system); (3) telephone contact with the study's Tobacco Coach (excluding the initial call after enrollment); (4) outpatient prescription for nicotine replacement, bupropion, or varenicline in the EHR; or (5) provision of nicotine replacement by the Quitline. Information was obtained from the EHR, research program records, practice-based tobacco counselor records, and the Quitline provider, National Jewish Health
Proportion of patients who are provided any evidence-based tobacco cessation treatment (defined below), comparing External Community Referral vs. Usual Care | 6 months
  Treatment defined as above
Proportion of patients who are provided any evidence-based tobacco cessation treatment (defined below), comparing Internal Care Coordination vs. External Community Referral | 6 months
  Treatment defined as above
Proportion of patients reporting cigarette abstinence for the past 7 days (point-prevalence abstinence measure) | 6 months
  Proportion of patients who report that they have not smoked a cigarette in the past 7 days on a telephone survey (point-prevalence abstinence measure)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Rigotti, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalkhoran S, Inman EM, Kelley JHK, Ashburner JM, Rigotti NA. Proactive Population Health Strategy to Offer Tobacco Dependence Treatment to Smokers in a Primary Care Practice Network. J Gen Intern Med. 2019 Aug;34(8):1571-1577. doi: 10.1007/s11606-019-05079-3. Epub 2019 Jun 13. PMID 31197730